CLINICAL TRIAL: NCT00246324
Title: An Open Label Trial of Safety and Efficacy of Combination Therapy With Interferon-B-1a and Oral Doxycycline in Patients With Relapsing-remitting Multiple Sclerosis (RRMS)
Brief Title: Safety and Efficacy Study of Doxycycline in Combination With Interferon-B-1a to Treat Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H04-090
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Interferon beta 1a, oral doxycycline
  Interventions: Drug: Interferon beta 1a, oral doxycycline

INTERVENTIONS:
Drug: Interferon beta 1a, oral doxycycline — Patients took intramuscular interferon beta 1a, 30 micrograms, for 3 months then added oral doxycycline, 100 daily with the interferon for 4 months.
  Other Names: Avonex

SUMMARY:
To evaluate the efficacy, safety, and tolerability of combination therapy with intramuscular interferon beta-1a and oral doxycycline, a potent inhibitor of matrix metalloproteinases, in patients with relapsing remitting multiple sclerosis (RRMS) having breakthrough disease activity.

DETAILED DESCRIPTION:
Eligible individuals were evaluated monthly for 3 months while taking intramuscular interferon beta-1a, 30 micrograms weekly, then monthly for 4 months while receiving intramuscular interferon beta-1a, 30 micrograms and oral doxycycline, 100 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* Relapsing-Remitting Multiple Sclerosis (RRMS)
* Avonex therapy for 6 months prior continuous
* annualized relapse rate >2 during Avonex therapy
* most recent relapse within 60 days of baseline
* entry Expanded Disability Status Scale (EDSS) 1.5-4.5
* one or more gadolinium (Gd+) MRI lesions on a baseline MRI
* no history of immune modulator or immunosuppressant therapy used in combination with Avonex (other then GSC administer for clinical relapses)
* not participating in any other study of ms therapeutics
* Serum neutralizing antibodies (NABs) titer to Avonex <20

Exclusion Criteria:

* Medical or Psychiatric conditions that will affect patients ability to provide informed consent
* inability to undergo MRI
* clinically serious medical conditions or significantly abnormal labs
* no use of these medications or procedures within six months prior to study:

  *monoclonal antibodies,total lymphoid radiation,systemic steroids,cytotoxic or immunosuppressive medications such as mitoxantrone or cyclophosphamide or any other investigational drugs
* Interferon neutralizing antibody titers >20
* no breast feeding or pregnant
* no patients with any systemic illness,psychiatric condition or other disorder that would concern safety of patient to complete procedures of protocol
* abnormal blood test
* clinically significant abnormality on chest x-ray (CXR)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-12; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Minagar, MD, Principal Investigator — LSU Health Sciences Center -Shreveport
Locations (1):
- LSU Health Sciences Center Shreveport, Shreveport, Louisiana, United States

REFERENCES:
- [Result] Minagar A, Alexander JS, Schwendimann RN, Kelley RE, Gonzalez-Toledo E, Jimenez JJ, Mauro L, Jy W, Smith SJ. Combination therapy with interferon beta-1a and doxycycline in multiple sclerosis: an open-label trial. Arch Neurol. 2008 Feb;65(2):199-204. doi: 10.1001/archneurol.2007.41. Epub 2007 Dec 10. PMID 18071030

RESULTS

PARTICIPANT FLOW:
Groups:
- Inteferon, Then Interferon With Doxycycline: Men and women with RRMS who had received interferon beta-1a intramuscularly for at least six months and were experiencing breakthrough disease activity with the most recent relapse within 60 days of study entry.
Period: Overall Study
Arm/Group | Inteferon, Then Interferon With Doxycycline
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Inteferon, Then Interferon With Doxycycline
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Gadolinium-enhancing (Gd+)Lesion Number Change.
Description: Before treatment is the number of lesions per image from months -3, -2, -1, and 0. During treatment is the number of lesions from months 1,2, and 3. The mean number of Gd+ lesions during each treatment period was calculated for each patient as the total number of Gd+ lesions observed across all images divided by the number of images. Hence, the mean number of Gd+ lesions per patient represents the number of lesions per MRI.
Time Frame: 8 months
Measure: Median (95% Confidence Interval); unit: Gd+ lesions
Arm/Group | Inteferon, Then Interferon With Doxycycline
Number analyzed (Participants) | 16
Gd+ lesions | 4.0 [0.7 to 16.7]

2. Secondary Outcome: Relapse Rates, Serum Matrix Metalloproteinase 9 Levels, Transendothelial Migration of Monocytes
Description: Only 1 patient relapsed. Correlations between decrease serum metalloproteinase 9 levels and enhancing lesion activity reduction. Transendothelial migration of monocytes was suppressed. Adverse effects were mild. No adverse synergistic effects of combination therapy.
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | Inteferon, Then Interferon With Doxycycline
Number analyzed (Participants) | 16
participants | 15

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 7 months
Arm/Group | Inteferon, Then Interferon With Doxycycline
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No